CLINICAL TRIAL: NCT02337283
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Doses of BI 425809 Tablets Given Orally Once Daily for 12 Days to Young and Elderly Healthy Male and Female Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Groups Phase I Study)(Part 1) and Comparison of Pharmacokinetics of a Single Oral Dose of BI 425809 After Oral Administration in the Morning Versus Oral Administration in the Evening in Young Healthy Male and Female Volunteers (Randomised, Two-sequence, Open, Two Period, Two-way Cross Over) (Part 2)
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Doses of BI 425809 Tablets for 12 Days to Young and Elderly Healthy Male and Female Volunteers and Comparison of Pharmacokinetics of a Single Oral Dose of BI 425809 (Morning Versus Evening)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1346.2; 2014-004390-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809

ARMS (7):
- BI 425809 very low dose - part I (Experimental): Part I only - very low dose tablet, oral administration with 240 ml water, over 14 days
  Interventions: Drug: BI 425809
- Placebo - part I (Placebo Comparator): Part I only - placebo tablet, oral administration with 240ml water, over 14 days
  Interventions: Drug: Placebo
- BI 425809 low dose - part I (Experimental): Part I - low dose tablet, oral administration with 240 ml water, over 14 days
  Interventions: Drug: BI 425809
- BI 425809 medium dose - part I (Experimental): Part I only - medium dose tablet, oral administration with 240 ml water, over 14 days
  Interventions: Drug: BI 425809
- BI 425809 high dose -part I (Experimental): Part I only - high dose tablet, oral administration with 240 ml water, over 14 days
  Interventions: Drug: BI 425809
- BI 425809 low dose - part II (Experimental): Part II - one low dose tablet on day 1 of visit 2 and 2a
  Interventions: Drug: BI 425809
- BI 425809 very high dose -part I (Experimental): Part I only - very high dose tablet, oral administration with 240 ml water, over 14 days
  Interventions: Drug: BI 425809

INTERVENTIONS:
Drug: BI 425809 — Tablets
  Other Names: Iclepertin
  Arms: BI 425809 high dose -part I; BI 425809 low dose - part I; BI 425809 low dose - part II; BI 425809 medium dose - part I; BI 425809 very high dose -part I; BI 425809 very low dose - part I
Drug: Placebo — Tablets
  Arms: Placebo - part I

SUMMARY:
The aim of the study is to investigate the safety, tolerability, and pharmacokinetics of multiple rising doses of BI 425809 tablets given orally once daily for 12 days to young and elderly healthy male and female volunteers and to compare single dose pharmacokinetics of BI 425809 given in the morning and in the evening.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects according to the investigator´s assessment, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* age of 18 to 50 years (incl.) for young healthy volunteers or age of 65 to 80 years (incl.) for elderly healthy volunteers
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and local legislation
* Female subjects who meet any of the following criteria:

  1. Surgically sterilised
  2. Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg in young subjects, and systolic blood pressure greater than 150 mmHg, diastolic blood pressure greater than 95 mmHg in elderly subjects, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* Further exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
frequency [N(%)] of subjects with drug related adverse events (AEs) | up to 25 days after first drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) only part II | up to 96 hours
Cmax (maximum measured concentration of the analyte in plasma) only part II | up to 96 hours

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after first dose
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) | up to 216 hours after last dose
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) | up to 216 hours after last dose
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) only part II | up to 96 hours
AUCt 0-24(area under the concentration-time curve of the analyte in plasma over a uniform dosing interval t after administration of the first dose) | up to 72 hours after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1346.2.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany

REFERENCES:
- [Derived] Moschetti V, Schlecker C, Wind S, Goetz S, Schmitt H, Schultz A, Liesenfeld KH, Wunderlich G, Desch M. Multiple Rising Doses of Oral BI 425809, a GlyT1 Inhibitor, in Young and Elderly Healthy Volunteers: A Randomised, Double-Blind, Phase I Study Investigating Safety and Pharmacokinetics. Clin Drug Investig. 2018 Aug;38(8):737-750. doi: 10.1007/s40261-018-0660-2. PMID 29846887